CLINICAL TRIAL: NCT01349803
Title: A Randomized, Double-blind, Parallel Group, 14-day, Multi-Center Study to Evaluate the Safety of PT003, PT005, PT001 and Foradil® Aerolizer® (12 µg, Open Label) as Evaluated by Holter Monitoring, in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: PT003 MDI Cardiovascular Safety Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT003003
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PT005 MDI (Experimental): PT005 MDI
  Interventions: Drug: PT005 MDI
- PT001 MDI (Experimental): PT001 MDI
  Interventions: Drug: PT001 MDI
- PT003 MDI (Experimental): PT003 MDI
  Interventions: Drug: PT003 MDI
- Formoterol Fumarate 12 μg (Foradil® Aerolizer®) (Active Comparator): Formoterol Fumarate 12 μg (Foradil® Aerolizer®)
  Interventions: Drug: Formoterol Fumarate 12 μg (Foradil® Aerolizer®)

INTERVENTIONS:
Drug: PT005 MDI — PT005 MDI administered as two puffs BID for 14 days
  Arms: PT005 MDI
Drug: PT001 MDI — PT001 MDI administered as two puffs BID for 14 days
  Arms: PT001 MDI
Drug: PT003 MDI — PT003 MDI administered as two puffs BID for 14 days
  Arms: PT003 MDI
Drug: Formoterol Fumarate 12 μg (Foradil® Aerolizer®) — Formoterol Fumarate 12 μg (Foradil® Aerolizer®) administered BID for 14 days
  Other Names: Foradil® Aerolizer®
  Arms: Formoterol Fumarate 12 μg (Foradil® Aerolizer®)

SUMMARY:
This study is primarily a safety study. The primary and secondary endpoints are based on 24-hour Holter monitor assessments obtained on Day 14 relative to baseline.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed written informed consent
* 40 - 80 years of age
* Clinical history of COPD with airflow limitation that is not fully reversible
* Females of non-child bearing potential or females of child bearing potential with negative pregnancy test; and acceptable contraceptive methods
* Current/former smokers with at least a 10 pack-year history of cigarette smoking
* A measured post- bronchodilator FEV1/FVC ratio of < or = 0.70
* A measured post- bronchodilator FEV1 > or = 750ml or 30% predicted and < or = 80% of predicted normal values
* Able to change COPD treatment as required by protocol
* Acceptable baseline (Visit 2) Holter monitor recording

Key Exclusion Criteria:

* Women who are pregnant or lactating
* Primary diagnosis of asthma
* Alpha-1 antitrypsin deficiency as the cause of COPD
* Active pulmonary diseases
* Prior lung volume reduction surgery
* Abnormal chest X-ray (or CT scan) not due to the presence of COPD
* Hospitalized due to poorly controlled COPD within 3 months of Screening
* Clinically significant medical conditions that preclude participation in the study (e.g. clinically significant abnormal ECG, uncontrolled hypertension, glaucoma, symptomatic prostatic hypertrophy)
* Cancer that has not been in complete remission for at least 5 years
* Treatment with investigational study drug or participation in another clinical trial or study within the last 30 days or 5 half lives
* Clinically significant abnormal findings during the baseline Holter recording
* Patients with a pacemaker or ICD/CRT/CRT_D devices

Other inclusion/exclusion criteria as defined by the protocol

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, M.D., Study Director — Pearl Therapeutics
Locations (20):
- United States (10):
  - Pearl Investigative Site, Glendale, Arizona
  - Pearl Investigative Site, Fullerton, California
  - Pearl Investigative Site, Los Angeles, California
  - Pearl Investigative Site, San Diego, California
  - Pearl Investigative Site, Pensacola, Florida
  - Pearl Investigative Site, Lafayette, Louisiana
  - Pearl Investigative Site, North Dartmouth, Massachusetts
  - Pearl Investigative Site, Livonia, Michigan
  - Pearl Investigative Site, Medford, Oregon
  - Pearl Investigative Site, San Antonio, Texas
- Australia (6):
  - Pearl Investigative Site, Glebe, New South Wales
  - Pearl Investigative Site, Caboolture, Queensland
  - Pearl Investigative Site, Dawpark, South Australia
  - Pearl Investigative Site, Toorak Gardens, South Australia
  - Pearl Investigative Site, Heidelberg, Victoria
  - Pearl Investigative Site, Nedlands, Western Australia
- New Zealand (4):
  - Pearl Investigative Site, Caversham, Dunedin
  - Pearl Investigative Site, Private Bag, Hamilton
  - Pearl Investigative Site, Tauranga, North Island
  - Pearl Investigative Site, Newtown, Wellington Region

REFERENCES:
- [Derived] Ferguson GT, Reisner C, Pearle J, DePetrillo P, Maes A, Martin UJ. Cardiovascular safety profile of a fixed-dose combination of glycopyrrolate and formoterol fumarate delivered via metered dose inhaler using co-suspension delivery technology. Pulm Pharmacol Ther. 2018 Apr;49:67-74. doi: 10.1016/j.pupt.2018.01.007. Epub 2018 Feb 4. PMID 29567116

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 15 sites throughout the US, Australia, and New Zealand from May 2011 - November 2011. Study participation was a maximum of 7 weeks.
Pre-assignment Details: Study was a multicenter, randomized, double-blind, parallel group, chronic dosing (14 days) study; each patient was randomized to receive 1 of 4 possible treatments over the course of a 14-day treatment period
Groups:
- FF MDI (PT005): FF MDI 9.6 mcg
- GP MDI (PT001): GP MDI 36 mcg
- GFF MDI (PT003): GFF MDI 36/9.6 mcg
- Foradil® Aerolizer®: Formoterol Fumarate 12 μg
Period: Overall Study
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Started | 60 | 58 | 60 | 59
Completed | 59 | 57 | 57 | 57
Not Completed | 1 | 1 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Protocol-specified criteria | 0 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population (all randomized subjects)
Groups:
- Total: Total of all reporting groups
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer® | Total
Number analyzed (Participants) | 60 | 58 | 60 | 59 | 237
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (8.13) | 63.3 (7.93) | 64.3 (7.38) | 64.1 (7.91) | 64.0 (7.80)
Gender [Count of Participants; unit: Participants]
  Female | 33 | 32 | 26 | 31 | 122
  Male | 27 | 26 | 34 | 28 | 115

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-Hour Mean Heart Rate Post-dose
Description: The primary safety objective of this study was to compare the change in mean heart rate averaged over 24 hours post-dose, following twice daily dosing over 14 days with PT003 MDI, PT005 MDI, PT001 MDI or Foradil Aerolizer compared to baseline in patients with moderate to severe chronic obstructive pulmonary disease (COPD).
Time Frame: 14 days
Population: Safety Holter Monitoring Population: a sub-set of the safety population that had at least 18 hours of Holter monitoring data at Screening and at Day 1 and/or Day 14. Exclusions from this population were identified prior to database lock and unblinding.
Measure: Least Squares Mean (95% Confidence Interval); unit: bpm
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 59 | 57 | 55 | 55
bpm | -0.19 [-1.38 to 1.00] | -1.84 [-3.05 to -0.63] | 0.40 [-0.84 to 1.63] | -0.09 [-1.32 to 1.15]

2. Secondary Outcome: Change From Baseline in Mean FEV1 Trough
Description: Trough FEV1 averaged over Day 7 and Day 14
Time Frame: Day 7 to Day 14
Population: MITT - patients from the ITT population who completed at least one evaluable FEV1 spirometry assessment for baseline (pre-dose on Day 1) and had an evaluable FEV1 spirometry assessment on at least one of the following: Day 7 pre-dose or Day 14 pre-dose (or both).
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 57 | 49 | 53 | 55
Liters | 0.091 [0.049 to 0.134] | 0.126 [0.080 to 0.172] | 0.251 [0.207 to 0.295] | 0.124 [0.081 to 0.167]

3. Secondary Outcome: Change From Baseline in 24-Hour Mean Heart Rate for Day 1 of Treatment
Description: The secondary objectives of the study was to further characterize cardiovascular safety parameters of all treatment groups including the maximum 24-hour heart rate, mean night-time and day-time heart rate, ventricular ectopic events, ventricular couplets, ventricular runs, the number of supraventricular runs, and sustained ventricular tachycardia (VT), supraventricular ectopic events, and other clinically relevant arrhythmias (such as atrial fibrillation).
Time Frame: 24 hours
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: bpm
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 60 | 58 | 57 | 57
bpm | 0.56 [-0.73 to 1.85] | -0.44 [-1.75 to 0.87] | 0.92 [-0.40 to 2.24] | 0.31 [-1.01 to 1.63]

4. Secondary Outcome: Change From Baseline in Daytime Mean Heart Rate
Description: as for outcome 3
Time Frame: Baseline, Day 1, and Day 14
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: bpm
Groups:
- FF MDI (PT005): FF MDI 9.6 mcg Day 1: N=59 Day 14: N=59
- GP MDI (PT001): GP MDI 36 mcg Day 1: N=58 Day 14: N=57
- GFF MDI (PT003): GFF MDI 36/9.6 mcg Day 1: N=57 Day 14: N=55
- Foradil® Aerolizer®: Formoterol Fumarate 12 μg Day 1: N=57 Day 14: N=55
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 59 | 58 | 57 | 57
bpm
  Day 1 | 0.00 [-1.40 to 1.40] | -0.52 [-1.93 to 0.90] | 0.16 [-1.27 to 1.58] | -0.17 [-1.60 to 1.25]
  Day 14 | -1.22 [-2.64 to 0.20] | -2.00 [-3.45 to -0.56] | -0.40 [-1.87 to 1.07] | -0.54 [-2.01 to 0.93]

5. Secondary Outcome: Change From Baseline in Night Time Mean Heart Rate
Description: as for outcome 3
Time Frame: Baseline, Day 1, and Day 14
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: bpm
Groups:
- FF MDI (PT005): FF MDI 9.6 mcg Day 1: N=59 Day 14: N=58
- GP MDI (PT001): GP MDI 36 mcg Day 1: N=57 Day 14: N=57
- GFF MDI (PT003): GFF MDI 36/9.6 mcg Day 1: N=55 Day 14: N=55
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 59 | 57 | 55 | 57
bpm
  Day 1 | 3.05 [1.63 to 4.47] | -0.54 [-1.99 to 0.90] | 2.95 [1.48 to 4.42] | 0.70 [-0.74 to 2.15]
  Day 14 | 0.04 [-1.94 to 2.03] | -0.88 [-2.89 to 1.12] | 0.11 [-1.93 to 2.15] | 1.05 [-0.99 to 3.09]

6. Secondary Outcome: Change From Baseline in 24-Hour Maximum Heart Rate
Description: as for outcome 3
Time Frame: Baseline, Day 1, and Day 14
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: bpm
Groups:
- FF MDI (PT005): FF MDI 9.6 mcg Day 1: N=60 Day 14: N=59
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 60 | 58 | 57 | 57
bpm
  Day 1 | -4.71 [-8.72 to -0.69] | -1.88 [-5.96 to 2.20] | -1.91 [-6.03 to 2.21] | 0.31 [-3.81 to 4.42]
  Day 14 | 0.75 [-3.46 to 4.97] | -2.21 [-6.50 to 2.07] | -0.06 [-4.42 to 4.31] | -1.13 [-5.49 to 3.23]

7. Secondary Outcome: Change From Baseline in 24-Hour Minimum Heart Rate
Description: as for outcome 3
Time Frame: Baseline, Day 1, and Day 14
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: bpm
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 60 | 58 | 57 | 57
bpm
  Day 1 | 0.05 [-1.19 to 1.29] | -0.03 [-1.30 to 1.23] | 0.50 [-0.78 to 1.78] | 0.45 [-0.82 to 1.72]
  Day 14 | -0.79 [-1.92 to 0.35] | -1.92 [-3.07 to -0.77] | -0.21 [-1.38 to 0.97] | 0.88 [-0.30 to 2.05]

8. Secondary Outcome: Change From Baseline in Number of Isolated Ventricular Events Recorded During 24-Hour Holter Monitoring
Description: as for outcome 3
Time Frame: Baseline, Day 1, and Day 14
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Ventricular events / hour
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 60 | 58 | 57 | 57
Ventricular events / hour
  Day 1 | 1.31 (1.605) [-0.25 to 0.24] | 0.56 (0.853) [-0.32 to 0.18] | 1.59 (1.879) [-0.19 to 0.31] | 0.45 (0.580) [-0.24 to 0.26]
  Day 14 | 3.09 (4.092) [-0.31 to 0.16] | 0.62 (1.088) [-0.50 to -0.03] | -0.10 (0.541) [-0.17 to 0.31] | -0.54 (0.424) [0.04 to 0.52]

9. Secondary Outcome: Change From Baseline in the Number of Ventricular Couplets Recorded During 24-Hour Holter Monitoring
Description: as for outcome 3
Time Frame: Baseline, Day 1, and Day 14
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Ventricular couplets / hour
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 60 | 58 | 57 | 57
Ventricular couplets / hour
  Day 1 | 0.09 (0.071) [-0.25 to 0.24] | 0.00 (0.005) [-0.32 to 0.18] | 0.00 (0.009) [-0.19 to 0.31] | 0.00 (0.005) [-0.24 to 0.26]
  Day 14 | 0.02 (0.021) [-0.31 to 0.16] | 0.00 (0.009) [-0.50 to -0.03] | -0.03 (0.033) [-0.17 to 0.31] | -0.01 (0.004) [0.04 to 0.52]

10. Secondary Outcome: Change From Baseline in the Number of Ventricular Runs Recorded During 24-Hour Holter Monitoring
Description: as for outcome 3
Time Frame: Baseline, Day 1, and Day 14
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Ventricular runs / hour
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 60 | 58 | 57 | 57
Ventricular runs / hour
  Day 1 | -0.003 (0.0024) [-0.25 to 0.24] | -0.001 (0.0017) [-0.32 to 0.18] | 0.001 (0.0019) [-0.19 to 0.31] | -0.003 (0.0040) [-0.24 to 0.26]
  Day 14 | -0.004 (0.0021) [-0.31 to 0.16] | 0.001 (0.0029) [-0.50 to -0.03] | 0.001 (0.0013) [-0.17 to 0.31] | -0.004 (0.0037) [0.04 to 0.52]

11. Secondary Outcome: Change From Baseline in the Number of Isolated Supraventricular Events Recorded During 24-Hour Holter Monitoring
Description: as for outcome 3
Time Frame: Baseline, Day 1, and Day 14
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Supraventricular events / hour
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 60 | 58 | 57 | 57
Supraventricular events / hour
  Day 1 | 7.72 (6.971) [-0.25 to 0.24] | 0.74 (0.804) [-0.32 to 0.18] | -4.55 (5.947) [-0.19 to 0.31] | 15.36 (16.359) [-0.24 to 0.26]
  Day 14 | 3.61 (5.179) [-0.31 to 0.16] | -9.29 (9.398) [-0.50 to -0.03] | 3.61 (5.179) [-0.17 to 0.31] | 5.81 (11.320) [0.04 to 0.52]

12. Secondary Outcome: Change From Baseline in the Number of Supraventricular Couplets Recorded During 24-Hour Holter Monitoring
Description: as for outcome 3
Time Frame: Baseline, Day 1, and Day 14
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Supraventricular couplets / hour
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 60 | 58 | 57 | 57
Supraventricular couplets / hour
  Day 1 | 0.03 (0.034) [-0.25 to 0.24] | 0.01 (0.021) [-0.32 to 0.18] | 0.05 (0.019) [-0.19 to 0.31] | 0.04 (0.065) [-0.24 to 0.26]
  Day 14 | 0.01 (0.025) [-0.31 to 0.16] | 0.00 (0.017) [-0.50 to -0.03] | 0.00 (0.018) [-0.17 to 0.31] | -0.02 (0.020) [0.04 to 0.52]

13. Secondary Outcome: Change From Baseline in the Number of Supraventricular Runs Recorded During 24-Hour Holter Monitoring
Description: as for outcome 3
Time Frame: Baseline, Day 1, and Day 14
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Supraventricular runs / hour
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 60 | 58 | 57 | 57
Supraventricular runs / hour
  Day 1 | 0.00 (0.014) [-0.25 to 0.24] | 0.02 (0.011) [-0.32 to 0.18] | 0.01 (0.011) [-0.19 to 0.31] | 0.01 (0.010) [-0.24 to 0.26]
  Day 14 | 0.01 (0.013) [-0.31 to 0.16] | 0.02 (0.015) [-0.50 to -0.03] | 0.00 (0.012) [-0.17 to 0.31] | 0.01 (0.014) [0.04 to 0.52]

14. Secondary Outcome: Change From Baseline in the Number of Bradycardia Episodes Recorded During 24-Hour Holter Monitoring
Description: as for outcome 3
Time Frame: Baseline, Day 1, and Day 14
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Bradycardia episodes / hour
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 60 | 58 | 57 | 57
Bradycardia episodes / hour
  Day 1 | -0.04 (0.139) [-0.25 to 0.24] | -0.02 (0.083) [-0.32 to 0.18] | 0.11 (0.193) [-0.19 to 0.31] | 0.03 (0.036) [-0.24 to 0.26]
  Day 14 | -0.02 (0.111) [-0.31 to 0.16] | 0.40 (0.210) [-0.50 to -0.03] | 0.27 (0.283) [-0.17 to 0.31] | 0.13 (0.132) [0.04 to 0.52]

15. Secondary Outcome: Change From Baseline in the Number of Tachycardia Episodes Recorded During 24-Hour Holter Monitoring
Description: as for outcome 3
Time Frame: Baseline, Day 1, and Day 14
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Tachycardia episodes / hour
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 60 | 58 | 57 | 57
Tachycardia episodes / hour
  Day 1 | -0.16 (0.170) [-0.25 to 0.24] | -0.24 (0.209) [-0.32 to 0.18] | -0.02 (0.160) [-0.19 to 0.31] | -0.09 (0.197) [-0.24 to 0.26]
  Day 14 | -0.23 (0.146) [-0.31 to 0.16] | -0.34 (0.229) [-0.50 to -0.03] | 0.22 (0.154) [-0.17 to 0.31] | -0.01 (0.206) [0.04 to 0.52]

16. Secondary Outcome: Mean Change From Baseline in QTcF Interval
Description: as for outcome 3
Time Frame: Baseline, Day 1, Day 7, and Day 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Number analyzed (Participants) | 60 | 58 | 60 | 59
msec
  Day 1: Post-dose 30 minutes | 1.53 (11.238) [-0.25 to 0.24] | 4.67 (12.548) [-0.32 to 0.18] | 3.27 (9.223) [-0.19 to 0.31] | 3.71 (9.816) [-0.24 to 0.26]
  Day 1: Post-dose 2 hours | 1.75 (13.861) [-0.31 to 0.16] | 3.57 (12.866) [-0.50 to -0.03] | 1.62 (13.785) [-0.17 to 0.31] | 5.25 (11.709) [0.04 to 0.52]
  Day 1: Post-dose 24 hours | -0.09 (13.309) | 1.23 (16.142) | -1.43 (12.724) | 0.36 (10.989)
  Day 7: Pre-dose | -1.80 (10.362) | 1.40 (14.713) | 1.06 (12.151) | 3.85 (12.599)
  Day 14: Pre-dose | -0.59 (12.523) | 1.79 (13.028) | -0.42 (11.910) | 1.53 (14.085)
  Day 14: Post-dose 30 minutes | 1.21 (13.350) | 4.10 (17.202) | 2.23 (13.194) | 1.20 (14.458)
  Day 14: Post-dose 2 hours | 0.44 (12.521) | 6.02 (16.774) | 5.01 (14.861) | 3.98 (14.135)
  Day 14: Post-dose 24 hours | -1.32 (12.738) | -0.05 (13.794) | -1.93 (11.269) | 1.44 (16.086)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and Serious Adverse Events (SAEs) were collected from the time the subject signs the informed consent form up to 14 days following the last dose of study drug.
Description: All patients who were randomized to a treatment, received at least one dose of the study treatment, and had any safety data after starting study treatment. A patient who used a study treatment, but took less than one full dose qualified for this population.
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Foradil® Aerolizer®
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/58 | 1/60 | 1/59
Other Adverse Events (participants affected / at risk) | 6/60 | 4/58 | 2/60 | 5/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FF MDI (PT005) (N=60) | GP MDI (PT001) (N=58) | GFF MDI (PT003) (N=60) | Foradil® Aerolizer® (N=59)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FF MDI (PT005) (N=60) | GP MDI (PT001) (N=58) | GFF MDI (PT003) (N=60) | Foradil® Aerolizer® (N=59)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Tremor (Nervous system disorders) | 4 (5) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.